CLINICAL TRIAL: NCT03079401
Title: Mesoblast Stem Cell Therapy for Patients With Single Ventricle and Borderline Left Ventricle
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sitaram Emani, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00020575
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Hypoplastic Left Heart Syndrome; Atrioventricular Canal
Keywords: biventricular conversion
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Endocardial Cushion Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Those randomized to the treatment arm will receive MPCs injected directly into the LV endocardium following clinical surgical maneuvers to recruit the LV (mitral valve repair, aortic valve repair, and/or resection of endocardial fibroelastosis) or BDG.
  MPCs will be delivered directly into the LV endocardium via a 23-25 gauge needle following completion of all surgical procedures. A total dose of 20 million cells will be delivered, divided evenly into ~11 injections of 50 µL each. The total volume is not to exceed 2.0 mL.
  Interventions: Biological: MPC; rexlemestrocel-L
- Control Arm (No Intervention): Those subjects randomized to the control arm will receive standard LV recruitment or BDG with no injection.

INTERVENTIONS:
Biological: MPC; rexlemestrocel-L — MPCs will be injected into the patient's myocardium during planned surgical procedures.
  Other Names: Allogeneic Mesenchymal Precursor Cell
  Arms: Treatment Arm

SUMMARY:
Patients under the age of 5, with a diagnosis of hypoplastic left heart syndrome (HLHS), unbalanced atrioventricular canal (uAVC), or borderline left heart who are undergoing staged LV recruitment following bidirectional Glenn (BDG) or undergoing BDG with plans for LV recruitment will be considered for enrollment in this study. Those patients enrolled in the study will be randomized to either the experimental arm or control arm of the study. Those patients randomized to the experimental arm will receive mesenchymal precursor cells (MPCs) injected directly into the LV endocardium during their LV recruitment or BDG procedure. Those patients randomized to the control arm will receive normal standard of care during their procedure with no injection of MPCs.

It is believed that injection of MPCs will help improve the chances of those patients with single ventricle or borderline left ventricle being converted to biventricular circulation which could improve quality of life and longevity over palliation.

DETAILED DESCRIPTION:
This is a prospective, single center, safety and feasibility, blinded, randomized trial to evaluate the use of MPCs in children with complex cardiac anatomy requiring surgical repair. Patients scheduled to undergo bidirectional Glenn (BDG) with future plans for LV recruitment, or patients with a history of BDG who are currently scheduled to undergo LV recruitment will be eligible.

Twenty-four subjects will be enrolled, 12 to the MPC treatment arm and 12 to the control arm following a 1:1 randomization schema. Randomization will be stratified according to surgeon to assure random distribution of subjects by surgeon. Families, the biostatistician, all clinical staff outside the operating room, and research staff completing data analysis will be blinded to randomization assignment. The PI, operating room staff, and research staff assisting with delivery will be unblinded to the randomization assignment. Families will be made aware of their randomization assignment once all subjects have completed their study Visit 4. Those randomized to the treatment arm will receive MPCs injected directly into the LV endocardium following clinical surgical maneuvers to recruit the LV (mitral valve repair, aortic valve repair, and/or resection of endocardial fibroelastosis) or BDG. Those subjects randomized to the control arm will receive standard LV recruitment or BDG with no injection.

All cardiac tissue acquired as part of a clinically indicated procedure will be collected on enrolled subjects. Most of the tissue sample will be analyzed at the time of collection (histology and H+E stain); the remainder will be banked for potential future testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of single ventricle palliation (Stage 1 palliation, PA band, or hybrid procedure) undergoing bidirectional Glenn (BDG) with simultaneous left ventricle (LV) recruitment procedures or those patients undergoing LV recruitment procedures will be considered for enrollment.

Exclusion Criteria:

* Patients with current or history of myocardial tumors
* Patients with aortic or mitral atresia
* Patients with a history of high grade ventricular arrhythmias
* Patients with a known allergy to dimethyl sulfoxide (DMSO)
* Patient has known allergy to mouse and/or cow products.
* Patient is prior recipient of stem cell therapy for cardiac repair.
* Patient has received treatment and/or is within an incomplete follow-up treatment of any investigational cell based therapy within 6 months prior to randomization.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Safety- Incidence of severe adverse events | 24 months
  Subjects will be SAE free for 24 months following injection of MPCs (in comparison of treatment arm to control arm.
Safety- Absence of PRA status change or local inflammation | 24 months
  Subjects will be free from Panel Reactive Antibody (PRA) status change for 24 months following injection of MPCs (in comparison of treatment arm to control arm). If there is a PRA of >5%, a donor specific antibody test will be completed,

SECONDARY OUTCOMES:
Efficacy- rate of biventricular conversion | 12 months
  Rate of those who are successfully converted to biventricular conversion in the treatment group compared to the control group.
Efficacy- improvement of LV end diastolic pressure | 12 months
  Rate of those who have improvement in these measurements in the treatment group compared to the control group.
Efficacy- improvement of LV mass/volume ratio | 12 months
  Rate of those who have improvement in these measurements in the treatment group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sitaram M Emani, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emani SM, del Nido PJ. Strategies to maintain biventricular circulation in patients with high-risk anatomy. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2013;16(1):37-42. doi: 10.1053/j.pcsu.2013.01.003. PMID 23561816
- [Background] Emani SM, McElhinney DB, Tworetzky W, Myers PO, Schroeder B, Zurakowski D, Pigula FA, Marx GR, Lock JE, del Nido PJ. Staged left ventricular recruitment after single-ventricle palliation in patients with borderline left heart hypoplasia. J Am Coll Cardiol. 2012 Nov 6;60(19):1966-74. doi: 10.1016/j.jacc.2012.07.041. Epub 2012 Oct 10. PMID 23062531
- [Background] Ascheim DD, Gelijns AC, Goldstein D, Moye LA, Smedira N, Lee S, Klodell CT, Szady A, Parides MK, Jeffries NO, Skerrett D, Taylor DA, Rame JE, Milano C, Rogers JG, Lynch J, Dewey T, Eichhorn E, Sun B, Feldman D, Simari R, O'Gara PT, Taddei-Peters WC, Miller MA, Naka Y, Bagiella E, Rose EA, Woo YJ. Mesenchymal precursor cells as adjunctive therapy in recipients of contemporary left ventricular assist devices. Circulation. 2014 Jun 3;129(22):2287-96. doi: 10.1161/CIRCULATIONAHA.113.007412. Epub 2014 Mar 28. PMID 24682346
- [Background] Psaltis PJ, Carbone A, Nelson AJ, Lau DH, Jantzen T, Manavis J, Williams K, Itescu S, Sanders P, Gronthos S, Zannettino AC, Worthley SG. Reparative effects of allogeneic mesenchymal precursor cells delivered transendocardially in experimental nonischemic cardiomyopathy. JACC Cardiovasc Interv. 2010 Sep;3(9):974-83. doi: 10.1016/j.jcin.2010.05.016. PMID 20850099